CLINICAL TRIAL: NCT07087925
Title: Comparison of Intravenous Haloperidol and Ondansetron Administered Intraoperatively in Reducing the Incidence of Postoperative Nausea and Vomiting (PONV) in Patients Undergoing Regional Anesthesia With Subarachnoid Block (RA-SAB)
Brief Title: Comparison of Haloperidol and Ondansetron in Reducing Postoperative Nausea and Vomiting in RA-SAB Patients
Acronym: HALO-PONV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rully Riyandika (Other)
Responsible Party: Sponsor-Investigator, Rully Riyandika, Sumatera Utara University, Universitas Sumatera Utara
Organization: Universitas Sumatera Utara (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HALO-ONDAN-PONV-RA-SAB; 1511/KEPK/USU/2024 (Other: Health Research Ethics Committee, Faculty of Medicine, Universitas Sumatera Utara)
Record Dates: First submitted 2025-07-16; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Postoperative Nausea and Vomiting (PONV); Subarachnoid Block; Spinal Anesthesia
Keywords: Haloperidol; Ondansetron; PONV; Regional Anesthesia; Subarachnoid Block; Spinal Anesthesia; Antiemetic Agents; Intraoperative Management; Postoperative Complications; Double-Blind Randomized Trial
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Postoperative Complications | interventions — Haloperidol; Ondansetron

STUDY DESIGN:
Intervention Model Description: A two-arm, randomized, double-blind, parallel assignment study comparing haloperidol and ondansetron administered intraoperatively to prevent PONV in patients undergoing subarachnoid block anesthesia.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind masking: Both participants and clinical team members, including data collectors and assessors, were unaware of the treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Haloperidol IV Group (Experimental): Participants in this arm received a single dose of intravenous haloperidol (1-2 mg) administered intraoperatively during surgery under subarachnoid block (RA-SAB). The goal was to evaluate its effectiveness in preventing postoperative nausea and vomiting (PONV). The administration was performed under blinded conditions, and patients were monitored for PONV occurrence and side effects for 24 hours postoperatively.
  Interventions: Drug: Haloperidol
- Ondansetron IV Group (Active Comparator): Participants in this arm received a single dose of intravenous ondansetron (4 mg) administered intraoperatively during surgery under subarachnoid block (RA-SAB). This group served as the active comparator to assess the relative effectiveness of ondansetron versus haloperidol in preventing PONV. Monitoring included assessment of PONV incidence and side effects for 24 hours postoperatively.
  Interventions: Drug: Ondansetron 4mg

INTERVENTIONS:
Drug: Haloperidol — A single dose of haloperidol (1-2 mg) was administered intravenously during the intraoperative period to patients undergoing surgery under subarachnoid block (RA-SAB). This intervention was designed to evaluate its effectiveness in preventing postoperative nausea and vomiting (PONV). Both patients and providers were blinded to the assignment.
  Arms: Haloperidol IV Group
Drug: Ondansetron 4mg — A single dose of ondansetron (4 mg) was administered intravenously during the intraoperative period to patients undergoing surgery under subarachnoid block (RA-SAB). This intervention served as the active comparator to haloperidol in evaluating the prevention of postoperative nausea and vomiting (PONV). The study was conducted in a double-blind manner.
  Arms: Ondansetron IV Group

SUMMARY:
This study aims to evaluate and compare the effectiveness of intravenous haloperidol and ondansetron in preventing postoperative nausea and vomiting (PONV) in patients undergoing surgery with subarachnoid block (spinal anesthesia). PONV is a common postoperative complication that can delay recovery, cause patient discomfort, and increase healthcare costs.

In this randomized, double-blind, prospective trial, eligible male patients aged 18-60 years undergoing elective surgeries under regional anesthesia were enrolled. Participants were assigned to receive either haloperidol or ondansetron during the intraoperative period. Both drugs are widely used antiemetic agents: haloperidol is a dopamine receptor antagonist, and ondansetron is a serotonin 5-HT3 receptor antagonist.

The primary objective was to assess the incidence of PONV within 24 hours after surgery. Results showed that haloperidol significantly reduced PONV incidence compared to ondansetron, with minimal adverse effects. The study suggests that intravenous haloperidol may be a cost-effective and well-tolerated alternative to ondansetron for PONV prevention in selected patients undergoing spinal anesthesia.

DETAILED DESCRIPTION:
Postoperative nausea and vomiting (PONV) remains one of the most common and distressing complications following surgery. Even with the use of regional anesthesia such as subarachnoid block (SAB), patients may still experience PONV, which affects recovery quality and increases healthcare burdens. Although antiemetic agents like ondansetron are commonly used, comparative studies evaluating alternative drugs such as haloperidol are limited, particularly in the context of spinal anesthesia.

This study was conducted to fill this gap by comparing the effectiveness of intravenous haloperidol and ondansetron in preventing PONV in patients undergoing surgery with subarachnoid block. The trial was carried out at RSUP H. Adam Malik Medan and Rumah Sakit Umum Haji Medan in Indonesia. A total of 40 male patients were recruited and randomly assigned into two groups to receive either intravenous haloperidol or ondansetron during the intraoperative period. The study design was double-blind, ensuring that both participants and medical personnel were unaware of the treatment allocations.

The primary outcome measured was the incidence of PONV within 24 hours after surgery. Data collection included patient demographics, APFEL risk scores, side effects (if any), and clinical observations. The haloperidol group had significantly fewer cases of PONV (2.5%) compared to the ondansetron group (30%). Additionally, both treatments were well tolerated with minimal adverse events. One case of mild sedation was noted in the haloperidol group, but no serious complications occurred in either group.

This study concludes that intravenous haloperidol is more effective than ondansetron in reducing PONV among male patients undergoing spinal anesthesia. Given its cost-effectiveness and favorable safety profile, haloperidol may be considered as an alternative antiemetic in clinical settings, particularly in resource-limited environments. However, further studies involving larger, gender-balanced populations are recommended to validate these findings and expand their generalizability.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged 18-60 years
* Undergoing elective surgery under regional anesthesia (Subarachnoid Block)
* Non-smokers
* Hemodynamically stable
* Surgical site involving gastrointestinal, pelvic, genital, perineal, or urologic regions
* Supine surgical position

Exclusion Criteria:

* Use of combined spinal and epidural anesthesia
* Known allergy to haloperidol or ondansetron
* Systemic infection, neuropathy, or coagulopathy
* Severe anxiety, psychiatric, or neuromuscular conditions
* Hormonal imbalances, gastritis, or pregnancy
* Conversion to general anesthesia due to block failure
* Intraoperative complications such as shock
* Abnormally prolonged surgery duration

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Incidence of Postoperative Nausea and Vomiting (PONV) within 24 Hours After Surgery | Within 24 hours postoperatively
  The occurrence of postoperative nausea and/or vomiting was assessed using a validated simplified PONV impact scale. Patients were monitored for symptoms such as nausea, vomiting, or dry retching within 24 hours after receiving either haloperidol or ondansetron. The outcome was recorded as binary (Yes/No).

CONTACTS AND LOCATIONS:
Locations (1):
- RSUP H. Adam Malik Medan, Medan, North Sumatra, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) related to primary and secondary outcomes-including incidence of PONV, sedation, and patient characteristics (age, BMI, APFEL score)-will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The IPD and supporting documents will be available starting 6 months after publication of the main study results and will remain accessible for 3 years thereafter.
Access Criteria: Qualified researchers may request access to the de-identified data and supporting materials for academic and non-commercial use. Requests must include a brief research proposal and data use agreement, and will be reviewed by the principal investigator. Approved users will receive data via secure email or institutional repository.